CLINICAL TRIAL: NCT03680391
Title: Effect of Early Posroperative Feeding on Gastrointestinal Function After Cesarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 41
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Post Operative Recovery
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early postoperative feeding: 103 patients will have early postoperative oral fluids and semisolid food after 6 hours of cesarean section irrespective to intestinal sounds ,flatus or stool passage
  Interventions: Procedure: Cesarean section
- Late postoperative feeding: 97 patient will start oral fluids 6 hours with no solid or semi solid until after passage of flatus or stool
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — Both groups cesarean section will be held with the same technique:
  * spinal anethesia
  * pfennenstiel imcision
  * lower segment cesarean section
  * suturing uterus in two layers while exterionezed
  * gentle manibulation
  * no towels in gutters will be used

SUMMARY:
Two hundred women were recruited, with 103 randomized to traditional feeding and 97 to early feeding and compare women satisfaction during discharge from hospital

DETAILED DESCRIPTION:
7. Study Methods

Population of study & disease condition :

Two hundred women were recruited, with 103 randomized to traditional feeding and 97 to early feeding and compare women satisfaction during discharge from hospital.

Inclusion criteria:

* Maternal age from 20 to 40
* Primigravida and previous one or two cesarean section
* Elective cesarean section
* regional anesthesia .singleton pregnancy.

Exclusion criteria:

* age below 20 years old or above 40 years old
* medical disorders as (hypertension, diabetes , liver or kidney diseases)
* complication during surgery as( bleeding, intestinal injury or urinary bladder injury ) .Emergency cesarean section .
* general anesthesia
* multiple pregnancy

Methodology in details:

1. all Women included in the study have undergo history taking and general examination
2. All patient in the study are randomized in two groups:

Group A:

103 patients will have early postoperative oral fluids and semisolid food after 6 hours of cesarean section irrespective to intestinal sounds ,flatus or stool passage

Group B:

97 patient will start oral fluids 6 hours with no solid or semi solid until after passage of flatus or stool 3_Both groups cesarean section will be held with the same technique:

* spinal anethesia
* pfennenstiel imcision
* lower segment cesarean section
* suturing uterus in two layers while exterionezed
* gentle manibulation
* no towels in gutters will be used 4_ comparison will be held between both groups according:
* postoperative intestinal sounds.
* postoperative nausea and vomiting
* postoprative abdominal distension
* postoperative pain
* postoperative ambulation
* postoperative ileus
* postoperative discharge time from hospital

ELIGIBILITY:
Inclusion Criteria:

* Maternal age from 20 to 40

  * Primigravida and previous one or two cesarean section
  * Elective cesarean section
  * regional anesthesia .singleton pregnancy.

Exclusion Criteria:

age below 20 years old or above 40 years old

* medical disorders as (hypertension, diabetes , liver or kidney diseases)
* complication during surgery as( bleeding, intestinal injury or urinary bladder injury ) .Emergency cesarean section .
* general anesthesia
* multiple pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Two hundred women were recruited, with 103 randomized to traditional feeding and 97 to early feeding and compare women satisfaction during discharge from hospital.
  1. all Women included in the study have undergo history taking and general examination
  2. All patient in the study are randomized in two groups:
  Group A:
  103 patients will have early postoperative oral fluids and semisolid food after 6 hours of cesarean section irrespective to intestinal sounds ,flatus or stool passage
  Group B:
  97 patient will start oral fluids 6 hours with no solid or semi solid until after passage of flatus or stool 3_Both groups cesarean section will be held with the same technique:
  * spinal anethesia
  * pfennenstiel imcision
  * lower segment cesarean section
  * suturing uterus in two layers while exterionezed
  * gentle manibulation
  * no towels in gutters will be used
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction before discharge from hospital | 2 days after the operation
  satisfaction score from 1 to 10 where 1 is totally non satisfied and 10 fully satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided